CLINICAL TRIAL: NCT06587841
Title: Noninvasive Spinal Cord Neuromodulation to Improve Lower Urinary Tract Function After Spinal Cord Injury in Ukrainian War Veterans
Brief Title: Noninvasive Spinal Cord Stimulation for Early SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Rivne Regional War Veterans Hospital, Spinal Cord Injury Rehabilitation Center (Unknown); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrei Krassioukov, MD, Professor in Physical Medicine and Rehabilitation, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-00284; CDMRP-SC230030 (Other: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2024-07-29; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Bowel Dysfunction; Sexual Dysfunction; Autonomic Dysfunction; Urologic Disorders
MeSH Terms: conditions — Spinal Cord Injuries; Intestinal Diseases; Sexual Dysfunction, Physiological; Primary Dysautonomias; Urologic Diseases

STUDY DESIGN:
Intervention Model Description: * Intervention Phase 1 (stimulation sessions) - 8 weeks: Participants will be randomized into one of two groups and be blinded to treatment assignment: Group 1 (treatment condition) will receive TSCS for 1 hour, 3 times/week; Group 2 (sham condition) will receive sham stimulation for 1 hour, 3 times/week.
  * Intervention Phase 2 (stimulation sessions) -8 weeks: Group 1 will continue to receive TSCS for 1 hour, 3 times/week, and Group 2 will switch from sham stimulation to TSCS for 1 hour, 3 times/week.
Who Masked: Participant
Masking Description: single-blinded, sham-controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Treatment (Experimental): TSCS at or between cervical spinal segment 5 (C5) and thoracic spinal segment 10 (T10) at Intervention Phases 1 and 2, 8 weeks each.
  Interventions: Device: Spinal COrd NEuromodulation™ (SCONE™) for transcutaneous spinal cord stimulation (TSCS)
- Group 2 Sham (Sham Comparator): TSCS at or between C5 and T10 at Intervention Phase 2; 8 weeks.
  Interventions: Device: Spinal COrd NEuromodulation™ (SCONE™) for transcutaneous spinal cord stimulation (TSCS)

INTERVENTIONS:
Device: Spinal COrd NEuromodulation™ (SCONE™) for transcutaneous spinal cord stimulation (TSCS) — The SCONE™ class II investigational device is a non-invasive central nervous system (CNS) stimulator (electrical continence device) designed to provide transcutaneous spinal cord stimulation for the improvement of symptoms of bladder dysfunction associated with centrally-mediated NLUTD.

SUMMARY:
The investigators are looking to determine the safety and efficacy of non-invasive transcutaneous spinal cord stimulation (TSCS) in promoting recovery of lower urinary tract (LUT), bowel, sexual, and cardiovascular function, as well as spasticity in individuals with subacute SCI (time since injury 3-6 months) and the impact on quality of life. The study will be conducted at two sites; site 1 in Canada and site 2 in the Ukraine. Up to 60 subjects will be enrolled; 10 adults at the ICORD, University of British Columbia (UBC), Vancouver, Canada site and 50 adults at the Rivne Regional War Veterans Hospital, Rivne, Ukraine. Eligible participants will be randomized (1:1 ratio) either to Group 1 (G1) or Group 2 (G2). G1 will receive therapeutic TSCS for 8 weeks (3 times per week; 1 hour per session) in conjunction with conventional rehabilitation (3-4 hours per day; 5 days per week). G2 will receive 8 weeks of sham stimulation in conjunction with conventional rehabilitation. After 8 weeks, G2 will cross over and receive therapeutic TSCS for 8 weeks, whereas G1 will continue to receive TSCS therapy for another 8 weeks, for a total of 16 weeks. Eligible participants enrolled into the study will attend fifty eight (58) visits for assessments, therapy, and follow-up. The expected duration of study participation for each participant will be 33 weeks.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of this clinical study is to investigate the safety and effectiveness of non-surgical transcutaneous spinal cord stimulation (TSCS) in helping with recovery of bladder function in individuals with SCI. Assessments: The immediate effects of TSCS (i.e., effects with stimulation on), long-term effects of TSCS, and the persisting effects of TSCS (i.e., any changes in function that are still present with stimulation off, after several weeks of using the stimulation regularly -pre versus post study comparison). This is a Phase II study. A Phase II study is undertaken after preliminary safety testing for a treatment.

Investigational Study Device:

The SCONE™ (Spinal COrd NEuromodulation) class II investigational device is a non-invasive central nervous system (CNS) stimulator (electrical continence device) designed to provide TSCS for the improvement of symptoms of bladder dysfunction associated with centrally-mediated NLUTD.

The SCONE™ device's primary mechanism of action is electrical stimulation delivered to the spinal cord through the skin. The device consists of an electrode connected by an electrical cable to a battery-powered pulse source and uses advanced waveforms to deliver electrical stimulation directly to the spinal cord neural networks associated with pelvic floor function with the aim to activate and retrain the neural circuits responsible for urinary bladder control.

Primary Objective:

To assess the effect of non-invasive TSCS on LUT function in people with sub-acute SCI following eight weeks of therapy in comparison to inactive sham control.

Secondary and Ancillary Objectives:

To assess the effect of non-invasive TSCS on bowel dysfunction, sexual dysfunctions, cardiovascular function, spasticity, and quality of life.

Specific Aim 1 - TSCS Mapping: To establish function-specific TSCS parameters and electrode placement to activate spinal neural circuits controlling LUT function in individuals with sub-acute SCI.

Primary Outcomes: Motor threshold (TSCS parameters) based on surface EMG for skeletal muscles innervated by motor neurons localized in the same spinal cord segments as neural circuits controlling LUT function [surface EMG of the EAS (surrogate for EUS)].

Hypothesis: In light of recent findings on the efficacy of spinal cord stimulation to improve LUT function, the optimal parameters for EMG responses (i.e., mapping) will be revealed during TSCS.

Specific Aim 2 -Effect of Real-Time TSCS: To test the safety and efficacy of real-time TSCS in improving LUT function in individuals with sub-acute SCI.

Primary Outcomes: Voiding efficiency of the bladder [surface EMG of the EAS (surrogate EUS)]; continuous cardiovascular monitoring for TSCS-dependent changes in BP i.e., adverse cardiovascular events such as AD.

Hypothesis: The investigators hypothesize that acute TSCS will reproducibly and safely improve voiding and storage functions in LUT and elicit pelvic floor EMG without any cardiovascular adverse events.

Specific Aim 3 - Effect of Long-Term TSCS: To investigate the efficacy of long-term TSCS in mitigating the NLUTD in the sub-acute period following SCI.

Primary Outcomes: Neurogenic Bladder Symptom Score (NBSS). Secondary outcomes: UDI and TNFBM. Ancillary Outcomes: Neurogenic Bowel Dysfunction (NBD) Score, sexual function screening tool, Sexual Health Inventory for Men (SHIM) Questionnaire, IIEF, FSFI, FSDS, 24hr ABPM, International Standards for Neurological Classification of SCI (ISNCSCI), Patient Health Questionnaire -9 (PHQ-9), PTSD Checklist for DSM-5 (PCL-5), WHO Quality of Life-BREF (WHOQOL-BREF), and modified Ashworth Score (MAS). Outcomes will be performed at baseline, 8- and 16-weeks post TSCS. Follow-up assessments will be performed 8 weeks after cessation of treatment to assess the persisting effects of TCS.

Hypothesis: Long-term TSCS will promote bladder/bowel voiding and storage functions as well as improvements in sexual function.

Specific Aim 4 - Effect of Delayed Onset TSCS: To investigate the efficacy of delayed long-term TSCS in mitigating NLUTD in the sub-acute period following SCI.

Primary Outcomes: NBSS. Secondary Outcomes: UDI and TNFBM. Ancillary Outcomes: NBD Score, sexual function screening tool, SHIM Questionnaire, IIEF, FSFI, FSDS, 24hr ABPM, ISNCSCI, PHQ-9, PCL-5, WHOQOL-BREF, and MAS. Outcomes will be performed at baseline, 8 weeks (sham) and 16 weeks (after 8 weeks of TSCS therapy). Follow-up assessments will be performed after cessation of TCS to assess the persisting effects of TSCS.

Hypothesis: Based on our promising preliminary findings in chronic SCI, the investigators hypothesize that even with delayed onset, TSCS will promote bladder/bowel voiding and storage functions, as well as boost sexual function.

Primary Efficacy Endpoint: Reduction in NBSS score by 10 points at 8 weeks of therapy.

Secondary Efficacy Endpoint: Mean improvement in voiding efficiency by at least 50%. Mean reduction in TNFBM by at least 50%.

RESEARCH DESIGN:

Overall Research Design:

The study will include sixty adults (19 - 65 years, n=50 in Ukraine and n=10 in Canada) with a sub-acute (time since injury of 3-6 months), motor-complete SCI [ASIA Impairment Scale (AIS) A or B] at spinal segments C5-T10, with documented impaired bladder function. The expected duration of study participation for each participant will be 33 weeks. Eligible Canadian participants enrolled into the study will attend 58 visits at ICORD.

Detailed Research Design:

The investigators propose a phase II, randomized, single-blinded, sham-controlled clinical trial to examine the effect of non-invasive TCS on LUT function in people with SCI. The investigators will include sixty adults (19 - 65 years, n=50 in Ukraine and n=10 in Canada) with a sub-acute (time since injury of 3-6 months), motor-complete SCI [AIS A or B] at spinal cord segments C5-T10, with documented impaired LUT function. Individuals with SCI will be recruited at Rivne Regional War Veterans Hospital for the Ukrainian site, and at ICORD for the Canadian site. The rationale for including the Canadian cohort (n=10) is to control for the environmental impact such as potential differences in intensity of sub-acute rehabilitation and severity of war-related psychological impact on functional recovery. Furthermore, participants will be instructed to adhere to established bowel and LUT routines and refrain from initiation of new medications for bowel and LUT management without notifying the Principal Investigator of this study.

Secondary and ancillary outcomes will include assessments of bowel function, sexual functions, cardiovascular function and spasticity. Group 1 (G1; n=25 in Ukraine and n=5 in Canada) will receive therapeutic TSCS for 8 weeks (3 times per week; 1 hour per session) in conjunction with conventional rehabilitation (3-4 hours per day; 5 days per week). G2 (n=25 in Ukraine and n=5 in Canada) will receive 8 weeks of sham stimulation in conjunction with conventional rehabilitation. After 8 weeks, G2 will switch to therapeutic TSCS for 8 weeks (i.e., delayed onset of TSCS). G1 will continue to receive TSCS therapy for another 8 weeks for a total of 16 weeks.

STATISTICAL PLAN & DATA ANALYSIS:

Short term changes in voiding efficiency and BP will be analyzed using paired t-tests (Aim 2). Primary and secondary outcome responder rates (i.e., proportion of participants realizing ≥10-point improvement from baseline in NBSS, 50% improvement in voiding efficiency, 50% reduction in TNFBM) will be analyzed using logistic regression (Aims 3 and 4). Primary, secondary, and ancillary outcomes will also be analyzed directly using mixed effects repeated measures models including fixed effects for treatment arm and country, and a random effect to account for nonindependence of repeated measurements within participants. Treatment-arm specific 95% confidence intervals will be constructed for all outcomes. Logistic, mixed effect models, and analysis of variance (ANOVA) (for short term changes in voiding efficiency and BP) will also incorporate interaction terms to examine differential effects associated with Ukraine-based vs Canada-based participants. Since the study is not powered for this assessment, interaction p<0.20 will be taken as evidence of possible differential effects and analyses limited to Ukraine-based participants only will be conducted separately. Interaction terms will also be included in mixed effects models to examine differential time trends between treatment arms (baseline to 8-week and 8-week to 16-week). Sham group 16-week outcomes will also be compared to experimental group 8-week outcomes (both having undergone 8 weeks of therapy to that point). Data transformations or nonparametric methods (e.g., Wilcoxon signed-rank test for paired data, Friedman test for nonparametric repeated measures) will be substituted in cases where distributional assumptions are not met. Analyses will include all participants completing each phase of the study; sensitivity analyses and multiple imputation will also be conducted as appropriate to examine the possible impact of attrition, which is expected to be low in this inpatient study. Analyses will not be corrected for multiple comparisons in view of the exploratory nature of many of the other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A participant must meet all of the following criteria in order to be eligible to participate:

  1. Age between 19 and 65 years at the time of consent
  2. Subacute SCI (time since injury 3-6months)
  3. ASIA Impairment Scale (AIS) A or B at spinal segments C5-T10
  4. Documented impaired LUT function
  5. Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

     i. Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit.

     ii. Women of childbearing potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence.
  6. Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment.
  7. Must provide informed consent.
  8. Agrees to comply with all planned visits and assessments, adhere with established bowel and LUT routines and refrain from initiation of new medications for bowel and LUT management without notifying the Principal Investigator of this study.

     Exclusion Criteria:
* A participant who meets any of the following criteria will be ineligible to participate:

  1. Clinically significant depression with thoughts of suicidal ideation (PHQ-9 total score above 20) or debilitating PTSD (PCL-5 total score above) or as judged by the investigator
  2. History of bladder augmentation or continent or incontinent urinary stoma or prior bladder surgery.
  3. Exhibits signs of lower motor neuron injury (i.e., concomitant conus medullaris/cauda equina injury).
  4. History of intradetrusor or intrasphincter onabotulinumtoxinA injections within 9 months of baseline visit.
  5. Concurrent use of any medication or treatment that in the opinion of the investigator interferes with study outcomes.
  6. Presence of cognitive impairments, social/psychological problems, or other comorbid conditions that, in the opinion of the Investigator, will preclude them from participation and completion of the study
  7. Presence of severe acute medical issues that interfere with testing (e.g., stage 3/4 pressure ulcers, uncontrolled diabetes).
  8. Contraindications for TSCS, such as:

     8.1. Implanted Cardiac pacemaker 8.2 Implanted metal in the trunk or spinal cord 8.3 Intrathecal delivery system (e.g., baclofen pump) 8.4 Implanted central or peripheral neuromodulator
  9. Medical condition that may put the participant at risk as determined by the investigator.
  10. Participation in or plans to participate in another research study that may interfere with the study endpoints.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Neurogenic Bladder Symptom Score (NBSS) | At baseline; At 8 weeks after treatment vs. sham; Following 16 weeks of stimulation; At 8 weeks after stopping stimulation
  Change in Neurogenic Bladder Symptom Score (NBSS) by 10-points at 8 weeks of therapy. The NBSS is a comprehensive and validated survey that quantifies symptoms of neurogenic lower urinary tract dysfunction (NLUTD). A minimum change of 5 points on the NBSS demonstrates clinically meaningful improvement for this patient population as established in the literature.

SECONDARY OUTCOMES:
Mean change in voiding efficacy by at least 50% | At baseline; At 8 weeks after treatment vs. sham; Following 16 weeks of stimulation; At 8 weeks after stopping stimulation
  Mean change in voiding efficacy by at least 50% related to bladder function as measured during urodynamic investigation (UDI).
  TSCS's efficacy assessment on lower urinary tract (LUT) function; The bladder will be prefilled without eliciting detrusor overactivity or autonomic dysreflexia (AD). Then, TSCS will be delivered in bursts (i.e., 60 seconds) interspersed with rest periods (i.e., 30 seconds) to improve voiding efficiency. It has been demonstrated that sacral neuromodulation can result in improvements in LUT function by over 50% compared to baseline.
Mean change in time needed for bowel movement (TNFBM) by at least 50% | At baseline; At 8 weeks after treatment vs. sham; Following 16 weeks of stimulation; At 8 weeks after stopping stimulation
  Mean change in time needed for bowel movement (TNFBM) by at least 50% related to bowel function as measured by the TNFBM.
  A conventional bowel routine (suppository use only) will be assessed three times over a one-week period. To assess and compare TNFBM, the time from 'suppository insertion' to 'when bowel evacuation is completed' at the individual's home will be recorded. Ninety-eight percent (98%) of individuals with SCI report at least one bowel issue, such as time needed for bowel management lasting up to 2 hrs., with over 60% reporting that bowel dysfunction adversely impacts their health related quality-of-life.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — The University of British Columbia, International Collaboration on Repair Discoveries (ICORD)
Locations (1):
- Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The research team plans to deposit final de-identified research data at a community-based repository for SCI research, such as Open Data Commons for SCI (https://odc-sci.org//). Research resources, including but not limited to, established stimulation parameter and recording equipment, will also be made available through material transfer agreement upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available upon full-text print publication in a peer-reviewed journal, for a duration of at least 10 years.
Access Criteria: Online access or e-mail request to the corresponding author from an established scientific investigator.

REFERENCES:
- [Background] Jackson AB, Dijkers M, Devivo MJ, Poczatek RB. A demographic profile of new traumatic spinal cord injuries: change and stability over 30 years. Arch Phys Med Rehabil. 2004 Nov;85(11):1740-8. doi: 10.1016/j.apmr.2004.04.035. PMID 15520968
- [Background] Dryden DM, Saunders LD, Jacobs P, Schopflocher DP, Rowe BH, May LA, Yiannakoulias N, Svenson LW, Voaklander DC. Direct health care costs after traumatic spinal cord injury. J Trauma. 2005 Aug;59(2):464-7. doi: 10.1097/01.ta.0000174732.90517.df. PMID 16294090
- [Background] Ackery A, Tator C, Krassioukov A. A global perspective on spinal cord injury epidemiology. J Neurotrauma. 2004 Oct;21(10):1355-70. doi: 10.1089/neu.2004.21.1355. PMID 15672627
- [Background] Hou S, Rabchevsky AG. Autonomic consequences of spinal cord injury. Compr Physiol. 2014 Oct;4(4):1419-53. doi: 10.1002/cphy.c130045. PMID 25428850
- [Background] Minervini G, Franco R, Marrapodi MM, Fiorillo L, Cervino G, Cicciu M. Post-traumatic stress, prevalence of temporomandibular disorders in war veterans: Systematic review with meta-analysis. J Oral Rehabil. 2023 Oct;50(10):1101-1109. doi: 10.1111/joor.13535. Epub 2023 Jun 23. PMID 37300526
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Wheeler TL; Bowel and Bladder Workshop Participants; de Groat W, Eisner K, Emmanuel A, French J, Grill W, Kennelly MJ, Krassioukov A, Gallo Santacruz B, Biering-Sorensen F, Kleitman N. Translating promising strategies for bowel and bladder management in spinal cord injury. Exp Neurol. 2018 Aug;306:169-176. doi: 10.1016/j.expneurol.2018.05.006. Epub 2018 May 10. PMID 29753647
- [Background] Strauss DJ, Devivo MJ, Paculdo DR, Shavelle RM. Trends in life expectancy after spinal cord injury. Arch Phys Med Rehabil. 2006 Aug;87(8):1079-85. doi: 10.1016/j.apmr.2006.04.022. PMID 16876553
- [Background] Garshick E, Kelley A, Cohen SA, Garrison A, Tun CG, Gagnon D, Brown R. A prospective assessment of mortality in chronic spinal cord injury. Spinal Cord. 2005 Jul;43(7):408-16. doi: 10.1038/sj.sc.3101729. PMID 15711609
- [Background] Squair JW, White BA, Bravo GI, Martin Ginis KA, Krassioukov AV. The Economic Burden of Autonomic Dysreflexia during Hospitalization for Individuals with Spinal Cord Injury. J Neurotrauma. 2016 Aug 1;33(15):1422-7. doi: 10.1089/neu.2015.4370. Epub 2016 Mar 22. PMID 27002855
- [Background] Hammell KR. Spinal cord injury rehabilitation research: patient priorities, current deficiencies and potential directions. Disabil Rehabil. 2010;32(14):1209-18. doi: 10.3109/09638280903420325. PMID 20131945
- [Background] Panicker JN, Fowler CJ, Kessler TM. Lower urinary tract dysfunction in the neurological patient: clinical assessment and management. Lancet Neurol. 2015 Jul;14(7):720-32. doi: 10.1016/S1474-4422(15)00070-8. PMID 26067125
- [Background] Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci. 2008 Jun;9(6):453-66. doi: 10.1038/nrn2401. PMID 18490916
- [Background] Pikov V, Gillis RA, Jasmin L, Wrathall JR. Assessment of lower urinary tract functional deficit in rats with contusive spinal cord injury. J Neurotrauma. 1998 May;15(5):375-86. doi: 10.1089/neu.1998.15.375. PMID 9605351
- [Background] David BT, Steward O. Deficits in bladder function following spinal cord injury vary depending on the level of the injury. Exp Neurol. 2010 Nov;226(1):128-35. doi: 10.1016/j.expneurol.2010.08.014. Epub 2010 Aug 14. PMID 20713043
- [Background] Consortium for Spinal Cord Medicine. Bladder management for adults with spinal cord injury: a clinical practice guideline for health-care providers. J Spinal Cord Med. 2006;29(5):527-73. No abstract available. PMID 17274492
- [Background] de Groat WC, Yoshimura N. Mechanisms underlying the recovery of lower urinary tract function following spinal cord injury. Prog Brain Res. 2006;152:59-84. doi: 10.1016/S0079-6123(05)52005-3. PMID 16198694
- [Background] Weld KJ, Dmochowski RR. Association of level of injury and bladder behavior in patients with post-traumatic spinal cord injury. Urology. 2000 Apr;55(4):490-4. doi: 10.1016/s0090-4295(99)00553-1. PMID 10736489
- [Background] Burns AS, St-Germain D, Connolly M, Delparte JJ, Guindon A, Hitzig SL, Craven BC. Phenomenological study of neurogenic bowel from the perspective of individuals living with spinal cord injury. Arch Phys Med Rehabil. 2015 Jan;96(1):49-55. doi: 10.1016/j.apmr.2014.07.417. Epub 2014 Aug 27. PMID 25172370
- [Background] Krassioukov A, Eng JJ, Claxton G, Sakakibara BM, Shum S. Neurogenic bowel management after spinal cord injury: a systematic review of the evidence. Spinal Cord. 2010 Oct;48(10):718-33. doi: 10.1038/sc.2010.14. Epub 2010 Mar 9. PMID 20212501
- [Background] Furness JB, Callaghan BP, Rivera LR, Cho HJ. The enteric nervous system and gastrointestinal innervation: integrated local and central control. Adv Exp Med Biol. 2014;817:39-71. doi: 10.1007/978-1-4939-0897-4_3. PMID 24997029
- [Background] Singh A, Tetreault L, Kalsi-Ryan S, Nouri A, Fehlings MG. Global prevalence and incidence of traumatic spinal cord injury. Clin Epidemiol. 2014 Sep 23;6:309-31. doi: 10.2147/CLEP.S68889. eCollection 2014. PMID 25278785
- [Background] Coggrave M, Norton C, Wilson-Barnett J. Management of neurogenic bowel dysfunction in the community after spinal cord injury: a postal survey in the United Kingdom. Spinal Cord. 2009 Apr;47(4):323-30; quiz 331-3. doi: 10.1038/sc.2008.137. Epub 2008 Nov 18. PMID 19015665
- [Background] Glickman S, Kamm MA. Bowel dysfunction in spinal-cord-injury patients. Lancet. 1996 Jun 15;347(9016):1651-3. doi: 10.1016/s0140-6736(96)91487-7. PMID 8642958
- [Background] Stone JM, Nino-Murcia M, Wolfe VA, Perkash I. Chronic gastrointestinal problems in spinal cord injury patients: a prospective analysis. Am J Gastroenterol. 1990 Sep;85(9):1114-9. PMID 2389723
- [Background] Lynch AC, Antony A, Dobbs BR, Frizelle FA. Bowel dysfunction following spinal cord injury. Spinal Cord. 2001 Apr;39(4):193-203. doi: 10.1038/sj.sc.3101119. PMID 11420734
- [Background] Lynch AC, Wong C, Anthony A, Dobbs BR, Frizelle FA. Bowel dysfunction following spinal cord injury: a description of bowel function in a spinal cord-injured population and comparison with age and gender matched controls. Spinal Cord. 2000 Dec;38(12):717-23. doi: 10.1038/sj.sc.3101058. PMID 11175370
- [Background] New PW. Secondary conditions in a community sample of people with spinal cord damage. J Spinal Cord Med. 2016 Nov;39(6):665-670. doi: 10.1080/10790268.2016.1138600. Epub 2016 Feb 23. PMID 26899984
- [Background] Simpson LA, Eng JJ, Hsieh JT, Wolfe DL; Spinal Cord Injury Rehabilitation Evidence Scire Research Team. The health and life priorities of individuals with spinal cord injury: a systematic review. J Neurotrauma. 2012 May 20;29(8):1548-55. doi: 10.1089/neu.2011.2226. Epub 2012 Apr 18. PMID 22320160
- [Background] Park SE, Elliott S, Noonan VK, Thorogood NP, Fallah N, Aludino A, Dvorak MF. Impact of bladder, bowel and sexual dysfunction on health status of people with thoracolumbar spinal cord injuries living in the community. J Spinal Cord Med. 2017 Sep;40(5):548-559. doi: 10.1080/10790268.2016.1213554. Epub 2016 Aug 31. PMID 27576584
- [Background] Alexander CJ, Sipski ML, Findley TW. Sexual activities, desire, and satisfaction in males pre- and post-spinal cord injury. Arch Sex Behav. 1993 Jun;22(3):217-28. doi: 10.1007/BF01541767. PMID 8494489
- [Background] Reitz A, Tobe V, Knapp PA, Schurch B. Impact of spinal cord injury on sexual health and quality of life. Int J Impot Res. 2004 Apr;16(2):167-74. doi: 10.1038/sj.ijir.3901193. PMID 14973522
- [Background] Sipski ML, Alexander CJ. Sexual activities, response and satisfaction in women pre- and post-spinal cord injury. Arch Phys Med Rehabil. 1993 Oct;74(10):1025-9. doi: 10.1016/0003-9993(93)90056-g. PMID 8215851
- [Background] Krassioukov A, Elliott S. Neural Control and Physiology of Sexual Function: Effect of Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2017 Winter;23(1):1-10. doi: 10.1310/sci2301-1. PMID 29339872
- [Background] Kandeel FR, Koussa VK, Swerdloff RS. Male sexual function and its disorders: physiology, pathophysiology, clinical investigation, and treatment. Endocr Rev. 2001 Jun;22(3):342-88. doi: 10.1210/edrv.22.3.0430. PMID 11399748
- [Background] Chen CH, Lin YC, Chiu LH, Chu YH, Ruan FF, Liu WM, Wang PH. Female sexual dysfunction: definition, classification, and debates. Taiwan J Obstet Gynecol. 2013 Mar;52(1):3-7. doi: 10.1016/j.tjog.2013.01.002. PMID 23548211
- [Background] Ibrahim E, Lynne CM, Brackett NL. Male fertility following spinal cord injury: an update. Andrology. 2016 Jan;4(1):13-26. doi: 10.1111/andr.12119. Epub 2015 Nov 4. PMID 26536656
- [Background] Giuliano F, Sanchez-Ramos A, Lochner-Ernst D, Del Popolo G, Cruz N, Leriche A, Lombardi G, Reichert S, Dahl P, Elion-Mboussa A, Casariego J. Efficacy and safety of tadalafil in men with erectile dysfunction following spinal cord injury. Arch Neurol. 2007 Nov;64(11):1584-92. doi: 10.1001/archneur.64.11.nct70001. Epub 2007 Sep 10. PMID 17846260
- [Background] Hess MJ, Hough S. Impact of spinal cord injury on sexuality: broad-based clinical practice intervention and practical application. J Spinal Cord Med. 2012 Jul;35(4):211-8. doi: 10.1179/2045772312Y.0000000025. PMID 22925747
- [Background] Curt A, Nitsche B, Rodic B, Schurch B, Dietz V. Assessment of autonomic dysreflexia in patients with spinal cord injury. J Neurol Neurosurg Psychiatry. 1997 May;62(5):473-7. doi: 10.1136/jnnp.62.5.473. PMID 9153603
- [Background] Karlsson AK. Autonomic dysreflexia. Spinal Cord. 1999 Jun;37(6):383-91. doi: 10.1038/sj.sc.3100867. PMID 10432257
- [Background] Sachdeva R, Nightingale TE, Krassioukov AV. The Blood Pressure Pendulum following Spinal Cord Injury: Implications for Vascular Cognitive Impairment. Int J Mol Sci. 2019 May 18;20(10):2464. doi: 10.3390/ijms20102464. PMID 31109053
- [Background] Hubli M, Gee CM, Krassioukov AV. Refined assessment of blood pressure instability after spinal cord injury. Am J Hypertens. 2015 Feb;28(2):173-81. doi: 10.1093/ajh/hpu122. Epub 2014 Jul 1. PMID 24990527
- [Background] Ho CP, Krassioukov AV. Autonomic dysreflexia and myocardial ischemia. Spinal Cord. 2010 Sep;48(9):714-5. doi: 10.1038/sc.2010.2. Epub 2010 Feb 2. PMID 20125109
- [Background] Eltorai I, Kim R, Vulpe M, Kasravi H, Ho W. Fatal cerebral hemorrhage due to autonomic dysreflexia in a tetraplegic patient: case report and review. Paraplegia. 1992 May;30(5):355-60. doi: 10.1038/sc.1992.82. PMID 1598177
- [Background] Wan D, Krassioukov AV. Life-threatening outcomes associated with autonomic dysreflexia: a clinical review. J Spinal Cord Med. 2014 Jan;37(1):2-10. doi: 10.1179/2045772313Y.0000000098. Epub 2013 Nov 26. PMID 24090418
- [Background] Phillips AA, Krassioukov AV. Contemporary Cardiovascular Concerns after Spinal Cord Injury: Mechanisms, Maladaptations, and Management. J Neurotrauma. 2015 Dec 15;32(24):1927-42. doi: 10.1089/neu.2015.3903. Epub 2015 Sep 1. PMID 25962761
- [Background] Kirshblum SC, House JG, O'connor KC. Silent autonomic dysreflexia during a routine bowel program in persons with traumatic spinal cord injury: a preliminary study. Arch Phys Med Rehabil. 2002 Dec;83(12):1774-6. doi: 10.1053/apmr.2002.36070. PMID 12474185
- [Background] Teasell RW, Arnold JM, Krassioukov A, Delaney GA. Cardiovascular consequences of loss of supraspinal control of the sympathetic nervous system after spinal cord injury. Arch Phys Med Rehabil. 2000 Apr;81(4):506-16. doi: 10.1053/mr.2000.3848. PMID 10768544
- [Background] Lee AHX, Phillips AA, Squair JW, Barak OF, Coombs GB, Ainslie PN, Sarafis ZK, Mijacika T, Vucina D, Dujic Z, Krassioukov AV. Alarming blood pressure changes during routine bladder emptying in a woman with cervical spinal cord injury. Spinal Cord Ser Cases. 2017 Dec 28;3:17101. doi: 10.1038/s41394-017-0022-y. eCollection 2017. PMID 29423304
- [Background] Liu N, Zhou MW, Biering-Sorensen F, Krassioukov AV. Cardiovascular response during urodynamics in individuals with spinal cord injury. Spinal Cord. 2017 Mar;55(3):279-284. doi: 10.1038/sc.2016.110. Epub 2016 Aug 2. PMID 27481090
- [Background] Faaborg PM, Christensen P, Krassioukov A, Laurberg S, Frandsen E, Krogh K. Autonomic dysreflexia during bowel evacuation procedures and bladder filling in subjects with spinal cord injury. Spinal Cord. 2014 Jun;52(6):494-8. doi: 10.1038/sc.2014.45. Epub 2014 Apr 29. PMID 24777164
- [Background] Krassioukov A, Warburton DE, Teasell R, Eng JJ; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of autonomic dysreflexia after spinal cord injury. Arch Phys Med Rehabil. 2009 Apr;90(4):682-95. doi: 10.1016/j.apmr.2008.10.017. PMID 19345787
- [Background] Pires PW, Dams Ramos CM, Matin N, Dorrance AM. The effects of hypertension on the cerebral circulation. Am J Physiol Heart Circ Physiol. 2013 Jun 15;304(12):H1598-614. doi: 10.1152/ajpheart.00490.2012. Epub 2013 Apr 12. PMID 23585139
- [Background] DeVivo MJ, Krause JS, Lammertse DP. Recent trends in mortality and causes of death among persons with spinal cord injury. Arch Phys Med Rehabil. 1999 Nov;80(11):1411-9. doi: 10.1016/s0003-9993(99)90252-6. PMID 10569435
- [Background] Myers J, Lee M, Kiratli J. Cardiovascular disease in spinal cord injury: an overview of prevalence, risk, evaluation, and management. Am J Phys Med Rehabil. 2007 Feb;86(2):142-52. doi: 10.1097/PHM.0b013e31802f0247. PMID 17251696
- [Background] Charlson F, van Ommeren M, Flaxman A, Cornett J, Whiteford H, Saxena S. New WHO prevalence estimates of mental disorders in conflict settings: a systematic review and meta-analysis. Lancet. 2019 Jul 20;394(10194):240-248. doi: 10.1016/S0140-6736(19)30934-1. Epub 2019 Jun 12. PMID 31200992
- [Background] Lehavot K, Goldberg SB, Chen JA, Katon JG, Glass JE, Fortney JC, Simpson TL, Schnurr PP. Do trauma type, stressful life events, and social support explain women veterans' high prevalence of PTSD? Soc Psychiatry Psychiatr Epidemiol. 2018 Sep;53(9):943-953. doi: 10.1007/s00127-018-1550-x. Epub 2018 Jun 23. PMID 29936598
- [Background] Williams R, Murray A. Prevalence of depression after spinal cord injury: a meta-analysis. Arch Phys Med Rehabil. 2015 Jan;96(1):133-40. doi: 10.1016/j.apmr.2014.08.016. Epub 2014 Sep 16. PMID 25220943
- [Background] Le J, Dorstyn D. Anxiety prevalence following spinal cord injury: a meta-analysis. Spinal Cord. 2016 Aug;54(8):626. doi: 10.1038/sc.2016.69. No abstract available. PMID 27492673
- [Background] Thuret S, Moon LD, Gage FH. Therapeutic interventions after spinal cord injury. Nat Rev Neurosci. 2006 Aug;7(8):628-43. doi: 10.1038/nrn1955. PMID 16858391
- [Background] Squair JW, West CR, Krassioukov AV. Neuroprotection, Plasticity Manipulation, and Regenerative Strategies to Improve Cardiovascular Function following Spinal Cord Injury. J Neurotrauma. 2015 May 1;32(9):609-21. doi: 10.1089/neu.2014.3743. Epub 2015 Apr 1. PMID 25582334
- [Background] Tator CH. Review of treatment trials in human spinal cord injury: issues, difficulties, and recommendations. Neurosurgery. 2006 Nov;59(5):957-82; discussion 982-7. doi: 10.1227/01.NEU.0000245591.16087.89. PMID 17143232
- [Background] Kwon BK, Hillyer J, Tetzlaff W. Translational research in spinal cord injury: a survey of opinion from the SCI community. J Neurotrauma. 2010 Jan;27(1):21-33. doi: 10.1089/neu.2009.1048. PMID 19751098
- [Background] Kwon BK, Okon E, Hillyer J, Mann C, Baptiste D, Weaver LC, Fehlings MG, Tetzlaff W. A systematic review of non-invasive pharmacologic neuroprotective treatments for acute spinal cord injury. J Neurotrauma. 2011 Aug;28(8):1545-88. doi: 10.1089/neu.2009.1149. Epub 2010 Apr 14. PMID 20146558
- [Background] Tetzlaff W, Okon EB, Karimi-Abdolrezaee S, Hill CE, Sparling JS, Plemel JR, Plunet WT, Tsai EC, Baptiste D, Smithson LJ, Kawaja MD, Fehlings MG, Kwon BK. A systematic review of cellular transplantation therapies for spinal cord injury. J Neurotrauma. 2011 Aug;28(8):1611-82. doi: 10.1089/neu.2009.1177. Epub 2010 Apr 20. PMID 20146557
- [Background] Silver J, Schwab ME, Popovich PG. Central nervous system regenerative failure: role of oligodendrocytes, astrocytes, and microglia. Cold Spring Harb Perspect Biol. 2014 Dec 4;7(3):a020602. doi: 10.1101/cshperspect.a020602. PMID 25475091
- [Background] Christison K, Walter M, Wyndaele JJM, Kennelly M, Kessler TM, Noonan VK, Fallah N, Krassioukov AV. Intermittent Catheterization: The Devil Is in the Details. J Neurotrauma. 2018 Apr 1;35(7):985-989. doi: 10.1089/neu.2017.5413. Epub 2018 Feb 1. PMID 29108476
- [Background] Esclarin De Ruz A, Garcia Leoni E, Herruzo Cabrera R. Epidemiology and risk factors for urinary tract infection in patients with spinal cord injury. J Urol. 2000 Oct;164(4):1285-9. PMID 10992382
- [Background] West DA, Cummings JM, Longo WE, Virgo KS, Johnson FE, Parra RO. Role of chronic catheterization in the development of bladder cancer in patients with spinal cord injury. Urology. 1999 Feb;53(2):292-7. doi: 10.1016/s0090-4295(98)00517-2. PMID 9933042
- [Background] Sugimura T, Arnold E, English S, Moore J. Chronic suprapubic catheterization in the management of patients with spinal cord injuries: analysis of upper and lower urinary tract complications. BJU Int. 2008 Jun;101(11):1396-400. doi: 10.1111/j.1464-410X.2007.07404.x. Epub 2008 Jan 8. PMID 18190633
- [Background] Wyndaele JJ, Madersbacher H, Kovindha A. Conservative treatment of the neuropathic bladder in spinal cord injured patients. Spinal Cord. 2001 Jun;39(6):294-300. doi: 10.1038/sj.sc.3101160. PMID 11438850
- [Background] Stohrer M, Blok B, Castro-Diaz D, Chartier-Kastler E, Del Popolo G, Kramer G, Pannek J, Radziszewski P, Wyndaele JJ. EAU guidelines on neurogenic lower urinary tract dysfunction. Eur Urol. 2009 Jul;56(1):81-8. doi: 10.1016/j.eururo.2009.04.028. Epub 2009 Apr 21. PMID 19403235
- [Background] Akkoc Y. Efficacy and safety of mirabegron for treatment of neurogenic detrusor overactivity in adults with spinal cord injury or multiple sclerosis: a systematic review. Spinal Cord. 2022 Oct;60(10):854-861. doi: 10.1038/s41393-022-00853-3. Epub 2022 Sep 9. PMID 36085413
- [Background] Walter M, Kran SL, Ramirez AL, Rapoport D, Nigro MK, Stothers L, Kavanagh A, Krassioukov AV. Intradetrusor OnabotulinumtoxinA Injections Ameliorate Autonomic Dysreflexia while Improving Lower Urinary Tract Function and Urinary Incontinence-Related Quality of Life in Individuals with Cervical and Upper Thoracic Spinal Cord Injury. J Neurotrauma. 2020 Sep 15;37(18):2023-2027. doi: 10.1089/neu.2020.7115. Epub 2020 Jul 23. PMID 32631152
- [Background] Sheel AW, Krassioukov AV, Inglis JT, Elliott SL. Autonomic dysreflexia during sperm retrieval in spinal cord injury: influence of lesion level and sildenafil citrate. J Appl Physiol (1985). 2005 Jul;99(1):53-8. doi: 10.1152/japplphysiol.00154.2005. Epub 2005 Mar 24. PMID 15790691
- [Background] Claydon VE, Elliott SL, Sheel AW, Krassioukov A. Cardiovascular responses to vibrostimulation for sperm retrieval in men with spinal cord injury. J Spinal Cord Med. 2006;29(3):207-16. doi: 10.1080/10790268.2006.11753876. PMID 16859224
- [Background] Fougere RJ, Currie KD, Nigro MK, Stothers L, Rapoport D, Krassioukov AV. Reduction in Bladder-Related Autonomic Dysreflexia after OnabotulinumtoxinA Treatment in Spinal Cord Injury. J Neurotrauma. 2016 Sep 15;33(18):1651-7. doi: 10.1089/neu.2015.4278. Epub 2016 Apr 13. PMID 26980078
- [Background] Squair JW, Phillips AA, Harmon M, Krassioukov AV. Emergency management of autonomic dysreflexia with neurologic complications. CMAJ. 2016 Oct 18;188(15):1100-1103. doi: 10.1503/cmaj.151311. Epub 2016 May 24. No abstract available. PMID 27221275
- [Background] Krassioukov A, Eng JJ, Warburton DE, Teasell R; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2009 May;90(5):876-85. doi: 10.1016/j.apmr.2009.01.009. PMID 19406310
- [Background] Phillips AA, Elliott SL, Zheng MM, Krassioukov AV. Selective alpha adrenergic antagonist reduces severity of transient hypertension during sexual stimulation after spinal cord injury. J Neurotrauma. 2015 Mar 15;32(6):392-6. doi: 10.1089/neu.2014.3590. Epub 2014 Dec 5. PMID 25093677
- [Background] Graham RM, Thornell IR, Gain JM, Bagnoli C, Oates HF, Stokes GS. Prazosin: the first-dose phenomenon. Br Med J. 1976 Nov 27;2(6047):1293-4. doi: 10.1136/bmj.2.6047.1293. No abstract available. PMID 793676
- [Background] Wecht JM, Rosado-Rivera D, Handrakis JP, Radulovic M, Bauman WA. Effects of midodrine hydrochloride on blood pressure and cerebral blood flow during orthostasis in persons with chronic tetraplegia. Arch Phys Med Rehabil. 2010 Sep;91(9):1429-35. doi: 10.1016/j.apmr.2010.06.017. PMID 20801263
- [Background] Nieshoff EC, Birk TJ, Birk CA, Hinderer SR, Yavuzer G. Double-blinded, placebo-controlled trial of midodrine for exercise performance enhancement in tetraplegia: a pilot study. J Spinal Cord Med. 2004;27(3):219-25. doi: 10.1080/10790268.2004.11753752. PMID 15478524
- [Background] James ND, McMahon SB, Field-Fote EC, Bradbury EJ. Neuromodulation in the restoration of function after spinal cord injury. Lancet Neurol. 2018 Oct;17(10):905-917. doi: 10.1016/S1474-4422(18)30287-4. Epub 2018 Sep 18. PMID 30264729
- [Background] Squair JW, Bjerkefors A, Inglis JT, Lam T, Carpenter MG. Cortical and vestibular stimulation reveal preserved descending motor pathways in individuals with motor-complete spinal cord injury. J Rehabil Med. 2016 Jul 18;48(7):589-96. doi: 10.2340/16501977-2101. PMID 27292455
- [Background] Gad PN, Roy RR, Zhong H, Lu DC, Gerasimenko YP, Edgerton VR. Initiation of bladder voiding with epidural stimulation in paralyzed, step trained rats. PLoS One. 2014 Sep 29;9(9):e108184. doi: 10.1371/journal.pone.0108184. eCollection 2014. PMID 25264607
- [Background] Abud EM, Ichiyama RM, Havton LA, Chang HH. Spinal stimulation of the upper lumbar spinal cord modulates urethral sphincter activity in rats after spinal cord injury. Am J Physiol Renal Physiol. 2015 May 1;308(9):F1032-40. doi: 10.1152/ajprenal.00573.2014. Epub 2015 Feb 18. PMID 25694482
- [Background] Meglio M, Cioni B, Amico ED, Ronzoni G, Rossi GF. Epidural spinal cord stimulation for the treatment of neurogenic bladder. Acta Neurochir (Wien). 1980;54(3-4):191-9. doi: 10.1007/BF01407085. PMID 6969533
- [Background] Herrity AN, Williams CS, Angeli CA, Harkema SJ, Hubscher CH. Lumbosacral spinal cord epidural stimulation improves voiding function after human spinal cord injury. Sci Rep. 2018 Jun 6;8(1):8688. doi: 10.1038/s41598-018-26602-2. PMID 29875362
- [Background] West CR, Phillips AA, Squair JW, Williams AM, Walter M, Lam T, Krassioukov AV. Association of Epidural Stimulation With Cardiovascular Function in an Individual With Spinal Cord Injury. JAMA Neurol. 2018 May 1;75(5):630-632. doi: 10.1001/jamaneurol.2017.5055. PMID 29459943
- [Background] Nightingale TE, Walter M, Williams AMM, Lam T, Krassioukov AV. Ergogenic effects of an epidural neuroprosthesis in one individual with spinal cord injury. Neurology. 2019 Feb 12;92(7):338-340. doi: 10.1212/WNL.0000000000006923. Epub 2019 Jan 11. No abstract available. PMID 30635485
- [Background] Zander HJ, Graham RD, Anaya CJ, Lempka SF. Anatomical and technical factors affecting the neural response to epidural spinal cord stimulation. J Neural Eng. 2020 Jun 12;17(3):036019. doi: 10.1088/1741-2552/ab8fc4. PMID 32365340
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Rattay F, Minassian K, Dimitrijevic MR. Epidural electrical stimulation of posterior structures of the human lumbosacral cord: 2. quantitative analysis by computer modeling. Spinal Cord. 2000 Aug;38(8):473-89. doi: 10.1038/sj.sc.3101039. PMID 10962608
- [Background] Ladenbauer J, Minassian K, Hofstoetter US, Dimitrijevic MR, Rattay F. Stimulation of the human lumbar spinal cord with implanted and surface electrodes: a computer simulation study. IEEE Trans Neural Syst Rehabil Eng. 2010 Dec;18(6):637-45. doi: 10.1109/TNSRE.2010.2054112. PMID 21138794
- [Background] Murg M, Binder H, Dimitrijevic MR. Epidural electric stimulation of posterior structures of the human lumbar spinal cord: 1. muscle twitches - a functional method to define the site of stimulation. Spinal Cord. 2000 Jul;38(7):394-402. doi: 10.1038/sj.sc.3101038. PMID 10962598
- [Background] Hofstoetter US, Freundl B, Binder H, Minassian K. Common neural structures activated by epidural and transcutaneous lumbar spinal cord stimulation: Elicitation of posterior root-muscle reflexes. PLoS One. 2018 Jan 30;13(1):e0192013. doi: 10.1371/journal.pone.0192013. eCollection 2018. PMID 29381748
- [Background] Phillips AA, Squair JW, Sayenko DG, Edgerton VR, Gerasimenko Y, Krassioukov AV. An Autonomic Neuroprosthesis: Noninvasive Electrical Spinal Cord Stimulation Restores Autonomic Cardiovascular Function in Individuals with Spinal Cord Injury. J Neurotrauma. 2018 Feb 1;35(3):446-451. doi: 10.1089/neu.2017.5082. Epub 2017 Nov 21. PMID 28967294
- [Background] Sachdeva R, Nightingale TE, Pawar K, Kalimullina T, Mesa A, Marwaha A, Williams AMM, Lam T, Krassioukov AV. Noninvasive Neuroprosthesis Promotes Cardiovascular Recovery After Spinal Cord Injury. Neurotherapeutics. 2021 Apr;18(2):1244-1256. doi: 10.1007/s13311-021-01034-5. Epub 2021 Mar 31. PMID 33791969
- [Background] Gad PN, Kreydin E, Zhong H, Latack K, Edgerton VR. Non-invasive Neuromodulation of Spinal Cord Restores Lower Urinary Tract Function After Paralysis. Front Neurosci. 2018 Jun 29;12:432. doi: 10.3389/fnins.2018.00432. eCollection 2018. PMID 30008661
- [Background] Inanici F, Brighton LN, Samejima S, Hofstetter CP, Moritz CT. Transcutaneous Spinal Cord Stimulation Restores Hand and Arm Function After Spinal Cord Injury. IEEE Trans Neural Syst Rehabil Eng. 2021;29:310-319. doi: 10.1109/TNSRE.2021.3049133. Epub 2021 Mar 2. PMID 33400652
- [Background] Aidoud A, Gana W, Poitau F, Debacq C, Leroy V, Nkodo JA, Poupin P, Angoulvant D, Fougere B. High Prevalence of Geriatric Conditions Among Older Adults With Cardiovascular Disease. J Am Heart Assoc. 2023 Jan 17;12(2):e026850. doi: 10.1161/JAHA.122.026850. Epub 2023 Jan 11. PMID 36628962
- [Background] Roehrborn CG. Benign prostatic hyperplasia: an overview. Rev Urol. 2005;7 Suppl 9(Suppl 9):S3-S14. PMID 16985902
- [Background] Krassioukov A, Linsenmeyer TA, Beck LA, Elliott S, Gorman P, Kirshblum S, Vogel L, Wecht J, Clay S. Evaluation and Management of Autonomic Dysreflexia and Other Autonomic Dysfunctions: Preventing the Highs and Lows: Management of Blood Pressure, Sweating, and Temperature Dysfunction. Top Spinal Cord Inj Rehabil. 2021 Spring;27(2):225-290. doi: 10.46292/sci2702-225. No abstract available. PMID 34108837
- [Background] Liu N, Fougere R, Zhou MW, Nigro MK, Krassioukov AV. Autonomic dysreflexia severity during urodynamics and cystoscopy in individuals with spinal cord injury. Spinal Cord. 2013 Nov;51(11):863-7. doi: 10.1038/sc.2013.113. Epub 2013 Sep 24. PMID 24060768
- [Background] Liu N, Zhou M, Biering-Sorensen F, Krassioukov AV. Iatrogenic urological triggers of autonomic dysreflexia: a systematic review. Spinal Cord. 2015 Jul;53(7):500-9. doi: 10.1038/sc.2015.39. Epub 2015 Mar 24. PMID 25800696
- [Background] Biering-Sorensen F, Craggs M, Kennelly M, Schick E, Wyndaele JJ. International lower urinary tract function basic spinal cord injury data set. Spinal Cord. 2008 May;46(5):325-30. doi: 10.1038/sj.sc.3102145. Epub 2007 Nov 27. PMID 18040278
- [Background] Kim JH, Rivas DA, Shenot PJ, Green B, Kennelly M, Erickson JR, O'Leary M, Yoshimura N, Chancellor MB. Intravesical resiniferatoxin for refractory detrusor hyperreflexia: a multicenter, blinded, randomized, placebo-controlled trial. J Spinal Cord Med. 2003 Winter;26(4):358-63. doi: 10.1080/10790268.2003.11753706. PMID 14992337
- [Background] Lombardi G, Del Popolo G, Cecconi F, Surrenti E, Macchiarella A. Clinical outcome of sacral neuromodulation in incomplete spinal cord-injured patients suffering from neurogenic bowel dysfunctions. Spinal Cord. 2010 Feb;48(2):154-9. doi: 10.1038/sc.2009.101. Epub 2009 Aug 11. PMID 19668257
- [Background] Hubli M, Krassioukov AV. Ambulatory blood pressure monitoring in spinal cord injury: clinical practicability. J Neurotrauma. 2014 May 1;31(9):789-97. doi: 10.1089/neu.2013.3148. Epub 2014 Jan 30. PMID 24175653
- [Background] Rupp R, Biering-Sorensen F, Burns SP, Graves DE, Guest J, Jones L, Read MS, Rodriguez GM, Schuld C, Tansey-Md KE, Walden K, Kirshblum S. International Standards for Neurological Classification of Spinal Cord Injury: Revised 2019. Top Spinal Cord Inj Rehabil. 2021 Spring;27(2):1-22. doi: 10.46292/sci2702-1. No abstract available. PMID 34108832
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Bombardier CH, Kalpakjian CZ, Graves DE, Dyer JR, Tate DG, Fann JR. Validity of the Patient Health Questionnaire-9 in assessing major depressive disorder during inpatient spinal cord injury rehabilitation. Arch Phys Med Rehabil. 2012 Oct;93(10):1838-45. doi: 10.1016/j.apmr.2012.04.019. Epub 2012 Apr 30. PMID 22555007
- [Background] Sakakibara BM, Miller WC, Orenczuk SG, Wolfe DL; SCIRE Research Team. A systematic review of depression and anxiety measures used with individuals with spinal cord injury. Spinal Cord. 2009 Dec;47(12):841-51. doi: 10.1038/sc.2009.93. Epub 2009 Jul 21. PMID 19621021
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Chang FS, Zhang Q, Xie HX, Wang HF, Yang YH, Gao Y, Fu CW, Chen G, Lu J. Preliminary validation study of the WHO quality of life (WHOQOL) scales for people with spinal cord injury in Mainland China. J Spinal Cord Med. 2022 Sep;45(5):710-719. doi: 10.1080/10790268.2020.1847563. Epub 2020 Dec 2. PMID 33263492
- [Background] Vahedi S. World Health Organization Quality-of-Life Scale (WHOQOL-BREF): Analyses of Their Item Response Theory Properties Based on the Graded Responses Model. Iran J Psychiatry. 2010 Fall;5(4):140-53. PMID 22952508
- [Background] Welk B, Morrow S, Madarasz W, Baverstock R, Macnab J, Sequeira K. The validity and reliability of the neurogenic bladder symptom score. J Urol. 2014 Aug;192(2):452-7. doi: 10.1016/j.juro.2014.01.027. Epub 2014 Feb 8. PMID 24518764
- [Background] Krogh K, Christensen P, Sabroe S, Laurberg S. Neurogenic bowel dysfunction score. Spinal Cord. 2006 Oct;44(10):625-31. doi: 10.1038/sj.sc.3101887. Epub 2005 Dec 13. PMID 16344850
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Barbonetti A, Cavallo F, Felzani G, Francavilla S, Francavilla F. Erectile dysfunction is the main determinant of psychological distress in men with spinal cord injury. J Sex Med. 2012 Mar;9(3):830-6. doi: 10.1111/j.1743-6109.2011.02599.x. Epub 2011 Dec 21. PMID 22188659
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Derogatis LR, Rosen R, Leiblum S, Burnett A, Heiman J. The Female Sexual Distress Scale (FSDS): initial validation of a standardized scale for assessment of sexually related personal distress in women. J Sex Marital Ther. 2002 Jul-Sep;28(4):317-30. doi: 10.1080/00926230290001448. PMID 12082670
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Welk B, Lenherr S, Elliott S, Stoffel J, Gomes CM, de Bessa J, Cintra LKL, Myers JB; Neurogenic Bladder Research Group. The creation and validation of a short form of the Neurogenic Bladder Symptom Score. Neurourol Urodyn. 2020 Apr;39(4):1162-1169. doi: 10.1002/nau.24336. Epub 2020 Mar 20. PMID 32196732
- [Background] Welk B, Lenherr S, Elliott S, Stoffel J, Presson AP, Zhang C, Myers JB. The Neurogenic Bladder Symptom Score (NBSS): a secondary assessment of its validity, reliability among people with a spinal cord injury. Spinal Cord. 2018 Mar;56(3):259-264. doi: 10.1038/s41393-017-0028-0. Epub 2017 Nov 29. PMID 29184133
- [Background] Ashley EA, Laskin JJ, Olenik LM, Burnham R, Steadward RD, Cumming DC, Wheeler GD. Evidence of autonomic dysreflexia during functional electrical stimulation in individuals with spinal cord injuries. Paraplegia. 1993 Sep;31(9):593-605. doi: 10.1038/sc.1993.95. PMID 8247602
- [Background] Tawashy AE, Eng JJ, Krassioukov AV, Warburton DE, Ashe MC, Hung C. Screening and habituation of functional electrical stimulation-leg cycle ergometry for individuals with spinal cord injury: a pilot study. J Neurol Phys Ther. 2008 Dec;32(4):164-70. doi: 10.1097/NPT.0b013e31818de56f. PMID 19265757
- [Background] Samejima S, Shackleton C, Malik RN, Cao K, Bohorquez A, Nightingale TE, Sachdeva R, Krassioukov AV. Spinal Cord Stimulation Prevents Autonomic Dysreflexia in Individuals with Spinal Cord Injury: A Case Series. J Clin Med. 2023 Apr 16;12(8):2897. doi: 10.3390/jcm12082897. PMID 37109234
- [Background] Kreydin E, Zhong H, Latack K, Ye S, Edgerton VR, Gad P. Transcutaneous Electrical Spinal Cord Neuromodulator (TESCoN) Improves Symptoms of Overactive Bladder. Front Syst Neurosci. 2020 Feb 6;14:1. doi: 10.3389/fnsys.2020.00001. eCollection 2020. PMID 32116576
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677
- [Background] Alrashidi AA, Nightingale TE, Currie KD, Hubli M, MacDonald MJ, Hicks AL, Oh P, Craven BC, Krassioukov AV. Exercise Improves Cardiorespiratory Fitness, but Not Arterial Health, after Spinal Cord Injury: The CHOICES Trial. J Neurotrauma. 2021 Nov 1;38(21):3020-3029. doi: 10.1089/neu.2021.0071. Epub 2021 Sep 3. PMID 34314235
- [Background] Walter M, Ramirez AL, Lee AHX, Nightingale TE, Rapoport D, Kavanagh A, Krassioukov AV. Fesoterodine Ameliorates Autonomic Dysreflexia While Improving Lower Urinary Tract Function and Urinary Incontinence-Related Quality of Life in Individuals With Spinal Cord Injury: A Prospective Phase IIa Study. J Neurotrauma. 2023 May;40(9-10):1020-1025. doi: 10.1089/neu.2022.0333. Epub 2022 Oct 25. PMID 36178342
- [Background] Bryce TN, Budh CN, Cardenas DD, Dijkers M, Felix ER, Finnerup NB, Kennedy P, Lundeberg T, Richards JS, Rintala DH, Siddall P, Widerstrom-Noga E. Pain after spinal cord injury: an evidence-based review for clinical practice and research. Report of the National Institute on Disability and Rehabilitation Research Spinal Cord Injury Measures meeting. J Spinal Cord Med. 2007;30(5):421-40. doi: 10.1080/10790268.2007.11753405. PMID 18092558
- [Background] Cook KF, Dunn W, Griffith JW, Morrison MT, Tanquary J, Sabata D, Victorson D, Carey LM, Macdermid JC, Dudgeon BJ, Gershon RC. Pain assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S49-53. doi: 10.1212/WNL.0b013e3182872e80. PMID 23479545
- [Background] Widerstrom-Noga E, Biering-Sorensen F, Bryce TN, Cardenas DD, Finnerup NB, Jensen MP, Richards JS, Siddall PJ. The International Spinal Cord Injury Pain Basic Data Set (version 2.0). Spinal Cord. 2014 Apr;52(4):282-6. doi: 10.1038/sc.2014.4. Epub 2014 Jan 28. PMID 24469147